CLINICAL TRIAL: NCT06085014
Title: Clinical and Electrophysiological Predictors of Arrhythmic Recurrence in Patients With Paroxysmal Atrial Fibrillation Undergoing First Transcatheter Ablation Procedure of Atrial Fibrillation by Pulmonary Vein Isolation
Brief Title: Clinical and Electrophysiological Predictors of Arrhythmic Recurrence in Patients With Paroxysmal AF Undergoing First Ablation Procedure of AF by Pulmonary Vein Isolation
Acronym: PREDICTORS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Sponsor
Other Study IDs: CCM 1981
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation Paroxysmal
Keywords: pulmonary vein isolation; atrial fibrillation; catheter ablation; electroanatomical map
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: Patients with paroxysmal AF with clinical indication to first transcatheter ablation procedure of AF by pulmonary vein isolation
  Interventions: Other: Standard of care
- Retrospective cohort: Patients who underwent ablative procedure in the two years prior to the start of the study
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Standard of care — All patients will undergo, as clinically indicated, AF ablation by pulmonary vein isolation achievable by radiofrequency, cryoenergy, or electroporation. All patients will preliminarily undergo electroanatomic mapping of the atrium by CARTO/Navx/Rhythmia system indifferently. Patients will be given follow-up visits at 3-6-12 months, during which any arrhythmic recurrences will be assessed
  Groups: Prospective cohort
Other: Data collection — There's no patient involvement. Data of patients who underwent ablative procedures two years before the start of the study will be retrospectively analyzed
  Groups: Retrospective cohort

SUMMARY:
From the literature, the success rate (i.e., absence of AF recurrence) of ablation in cases of paroxysmal AF at one year changes between 70 and 85 percent. This rate is considered suboptimal. Currently there are no data that can assess which factors are predictive of recurrence both clinically and electrophysiologically. In particular, it is not known whether and to what extent the atrial substrate present under baseline conditions affects the success rate of the procedure and what relationships exist with other predictors such as age, sex, atrial size at echo, and duration of arrhythmia.

DETAILED DESCRIPTION:
This is a multicenter prospective and retrospective observational study aimed at examining the role of the left atrial substrate and other baseline clinical variables on the efficacy of transcatheter ablation in patients with paroxysmal atrial fibrillation (AF) who underwent pulmonary vein isolation regardless of the power source and balloon or "point by point" catheters used.

The study will evaluate whether there are baseline clinical or electrophysiological features that can predict the success of transcatheter atrial fibrillation ablation even before it is performed, so as to assess which patients may actually benefit, and which patients should instead undergo more extensive ablative procedures in conjunction with pulmonary vein isolation to achieve an optimal success rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for AF ablation
* Adequate anticoagulation therapy according to CHADs VASC

Exclusion Criteria:

* patients who had already undergo an AF ablation procedure
* Presence of intracavitary thrombus
* Ejection fraction <35%
* Pregnancy
* Hematologic contraindications to ionizing radiation exposure
* Congenital heart diseases
* Cardiac Surgery < 1month
* Uncontrolled heart failure
* Valvular disease
* Contraindications to general anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal AF with clinical indication to first transcatheter ablation procedure of AF by pulmonary vein isolation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Assess clinical and electrophysiological predictors of arrhythmic recurrence | through study completion, an average of 1 year
  Evaluate the role of atrial disease, assessed by baseline electroanatomic mapping, age, gender, echocardiographic data, years from first AF episode, in predicting AF recurrence after AF ablation.

SECONDARY OUTCOMES:
Evaluate acute and mid- to long-term efficacy, safety, and procedural timing of different technologies | through study completion, an average of 1 year
  Evaluate mid and long term efficacy, safety, procedural timing between Cryo ablation, Pulsed Field Ablation, Radio Frequency ablation, point by point or single shot ablation of paroxysmal atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Riva, MD, Principal Investigator — IRCCS Centro Cardiologico Monzino
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Universitaria delle Marche, Ancona
  - IRCCS Centro Cardiologico Monzino, Milan

REFERENCES:
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Verma A, Wazni OM, Marrouche NF, Martin DO, Kilicaslan F, Minor S, Schweikert RA, Saliba W, Cummings J, Burkhardt JD, Bhargava M, Belden WA, Abdul-Karim A, Natale A. Pre-existent left atrial scarring in patients undergoing pulmonary vein antrum isolation: an independent predictor of procedural failure. J Am Coll Cardiol. 2005 Jan 18;45(2):285-92. doi: 10.1016/j.jacc.2004.10.035. PMID 15653029
- [Background] Rolf S, Kircher S, Arya A, Eitel C, Sommer P, Richter S, Gaspar T, Bollmann A, Altmann D, Piedra C, Hindricks G, Piorkowski C. Tailored atrial substrate modification based on low-voltage areas in catheter ablation of atrial fibrillation. Circ Arrhythm Electrophysiol. 2014 Oct;7(5):825-33. doi: 10.1161/CIRCEP.113.001251. Epub 2014 Aug 23. PMID 25151631
- [Background] Tijskens M, Bergonti M, Spera F, Ascione C, Saenen J, Huybrechts W, Miljoen H, Riva S, Wittock A, Heidbuchel H, Tondo C, Sarkozy A. Etiology and Outcome of Catheter Ablation in Patients With Onset of Atrial Fibrillation <45 Years of Age. Am J Cardiol. 2022 Mar 1;166:45-52. doi: 10.1016/j.amjcard.2021.11.030. Epub 2021 Dec 24. PMID 34961604
- [Background] Vlachos K, Efremidis M, Letsas KP, Bazoukis G, Martin R, Kalafateli M, Lioni L, Georgopoulos S, Saplaouras A, Efremidis T, Liu T, Valkanas K, Karamichalakis N, Asvestas D, Sideris A. Low-voltage areas detected by high-density electroanatomical mapping predict recurrence after ablation for paroxysmal atrial fibrillation. J Cardiovasc Electrophysiol. 2017 Dec;28(12):1393-1402. doi: 10.1111/jce.13321. Epub 2017 Sep 8. PMID 28884923
- [Background] Kirstein B, Neudeck S, Gaspar T, Piorkowski J, Wechselberger S, Kronborg MB, Zedda A, Hankel A, El-Armouche A, Tomala J, Schmidt T, Mayer J, Wagner M, Ulbrich S, Pu L, Richter U, Huo Y, Piorkowski C. Left atrial fibrosis predicts left ventricular ejection fraction response after atrial fibrillation ablation in heart failure patients: the Fibrosis-HF Study. Europace. 2020 Dec 23;22(12):1812-1821. doi: 10.1093/europace/euaa179. PMID 32830233
- [Background] Bergonti M, Spera FR, Ferrero TG, Nsahlai M, Bonomi A, Tijskens M, Boris W, Saenen J, Huybrechts W, Miljoen H, Gonzalez-Juanatey JR, Martinez-Sande JL, Vandaele L, Wittock A, Heidbuchel H, Valderrabano M, Rodriguez-Manero M, Sarkozy A. Characterization of Atrial Substrate to Predict the Success of Pulmonary Vein Isolation: The Prospective, Multicenter MASH-AF II (Multipolar Atrial Substrate High Density Mapping in Atrial Fibrillation) Study. J Am Heart Assoc. 2023 Jan 3;12(1):e027795. doi: 10.1161/JAHA.122.027795. Epub 2022 Dec 24. PMID 36565183